CLINICAL TRIAL: NCT05089331
Title: Recovery and Outcomes From Stroke-Longitudinal Assessment With Neuroimaging
Brief Title: ROSE-Longitudinal Assessment With Neuroimaging
Acronym: ROSE-LAWN
Status: Recruiting | Type: Observational
Sponsor: State University of New York at Buffalo (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); University of Maryland, Baltimore (Other); Duke University (Other); Columbia University (Other); University of Illinois at Chicago (Other); Baptist Health, Louisville (Other); The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Daniel Woo, M.D.,M.S., Professor, State University of New York at Buffalo
Other Study IDs: R01NS120493-02 (NIH); R01NS120493 (NIH)
Record Dates: First submitted 2021-10-11; First posted 2021-10-22 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Intracerebral Hemorrhage
Keywords: Hemorrhagic Stroke, Intracerebral; Intracerebral Hemorrhage; Outcomes after Stroke; Intracerebral hematoma
MeSH Terms: conditions — Cerebral Hemorrhage; Hemorrhagic Stroke

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, DNA, RNA and Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants will be recruited from the GERFHS/ROSE Study: Participants will be recruited who have had a hemorrhagic stroke and have been enrolled into the Genetic and Environmental Risk Factors for Hemorrhagic Stroke Study/Recovery and Outcomes from Stroke study, who live in the area of University of Cincinnati, University of Maryland, Duke University, Columbia University and University of Chicago Illinois, Baptist Health Louisville and Houston Methodist. The participant's age must be18 years or greater. The participant or legal representative must be able to provide informed consent, and the racial/ethnic category of participants should be Caucasian, African American or Hispanic.

SUMMARY:
The investigators will perform follow-up on 250 of 500 cases recruited into the ROSE study of cases with deep and lobar intracerebral hemorrhage to perform advanced neuroimaging at 12-24 months post stroke, and evaluations of motor and cognitive function at baseline, 6 months after baseline, and 12 months after baseline to determine predictors of recovery, progressive cognitive or functional impairment. The investigators propose to leverage the recruitment, DNA, RNA-seq and baseline advanced neuroimaging cohort of ROSE to obtain long-term neuroimaging and identical assessments longitudinally to address critical questions regarding the progressive decline of patients 12 to 24 months post intracerebral hemorrhage (ICH) with long term cognitive follow-up to 36 months on average. This proposal would represent the largest, and longest advanced neuroimaging and RNA-sequencing evaluation after ICH to date.

DETAILED DESCRIPTION:
The investigators propose to leverage the recruitment, DNA, RNA-seq and baseline advanced neuroimaging cohort of ROSE to obtain long-term neuroimaging and identical assessments longitudinally to address critical questions regarding the progressive decline of patients 12 to 24 months post ICH with long term cognitive follow-up to 36 months on average. This proposal would represent the largest, and longest advanced neuroimaging and RNA-sequencing evaluation after ICH to date.

Specific Aim #1: Determine if progressive cognitive impairment correlates with an increase in established markers of cerebral small vessel disease(CSVD) and cerebral amyloid angiopathy(CAA) (white matter disease, siderosis and microbleeds).

Hypothesis #1: Incidence of progressive cognitive impairment after ICH will be associated with an increase in total burden of small vessel disease (including white matter disease (WMD), microbleeds or siderosis, perivascular spaces, lacunar infarcts and atrophy).

Specific Aim #2: Determine if inflammation as measured by RNA-sequencing markers of inflammation correlates with progressive cognitive impairment.

Hypothesis #2: Interleukin-8 related inflammation will be associated with incidence of cognitive impairment.

Specific Aim #3: In this exploratory aim, we seek to identify novel neuroimaging markers associated with progressive cognitive decline.

Exploratory Hypothesis #3: Contralateral hemispheric diffusion tensor imaging (DTI) measures and cortical to cortical tract integrity will decline in association with progressive cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or greater, fulfillment of the criteria for Deep, Subcortical or Lobar Intracerebral Hemorrhage
* No evidence of trauma, vascular malformation or aneurysm, or brain tumor as a cause of ICH.
* Ability of the patient or legal representative to provide informed consent

Exclusion Criteria:

* Brainstem or Cerebellar ICH
* Patients Severely Affected by the ICH, Early Mortality, Hospice, or Withdraw of Care NOT eligible for ROS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants already enrolled in Genetic and Environmental Risk Factors for Hemorrhagic Stroke/Recovery and Outcomes from Stroke (GERFHS/ROSE) study
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-09-30 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Determination of whether progressive cognitive impairment correlates with CVD and AA markers | Ongoing/completed by September 2024
  Each subject has a baseline # Tesla (3T) MRI with DTI along with blinded central measurement of cerebral small vessel disease parameters. The current proposal is specifically designed to address these potential hypotheses by a comprehensive evaluation of detailed neurocognitive evaluations, baseline and long-term follow-up neuroimaging markers of CSVD and CAA as well as RNA sequencing of serum leukocytes for markers of inflammation.
Determination of whether inflammation as measured by RNA-sequencing markers of inflammation correlates with progressive cognitive impairment | Ongoing/completed by September 2024
  The current proposal is specifically designed to address these potential hypotheses by a comprehensive evaluation of detailed neurocognitive evaluations, baseline and long-term follow-up neuroimaging markers of CSVD and CAA as well as RNA sequencing of serum leukocytes for markers of inflammation. If the occurrence of progressive cognitive decline is caused by inflammation from the ICH itself, those with cognitive decline should have chronically increased expression of inflammation compared to those without cognitive decline, where inflammatory markers normalize. Our preliminary data suggests a role of interleukin-8 as increased in expression after ICH.

OTHER OUTCOMES:
Identification of neuroimaging markers associated with progressive cognitive decline | Ongoing/completed by September 2024
  The baseline and planned follow-up MRI include tractography to assess cortical to cortical tract integrity as well as inflammatory microstructural quantitative measurements. The follow-up MR tractography biomarkers will be compared to the acute/baseline MRI to determine if deterioration (particularly the contralateral hemisphere) correlates with progressive cognitive impairment. If the progressive deterioration in survivors of ICH is global, the contralateral hemisphere should also demonstrate progressive neuroimaging markers of deterioration.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Woo, MD, MS, Principal Investigator — State University of New York at Buffalo
Locations (7):
- United States (7):
  - University of Illinois Chicago, Chicago, Illinois
  - Baptist Health Louisville, Louisville, Kentucky
  - University of Maryland, Baltimore, Maryland
  - Columbia University, New York, New York
  - Duke University, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Houston Methodist, Houston, Texas

IPD SHARING:
Plan to Share IPD: No